CLINICAL TRIAL: NCT02151071
Title: A Pilot Study to Evaluate Molecular Imaging Using a BetaScope and a Specimen Analyser for Determining Margin and Lymph Node Status During Breast Conserving Surgery in Women With Breast Cancer
Brief Title: The Breast Surgery EnLight and LightPath Imaging System Study
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lightpoint Medical Limited (Industry)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other); King's College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LPM-002
Record Dates: First submitted 2014-05-27; First posted 2014-05-30 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Breast Neoplasms
Keywords: Breast Cancer; Mastectomy, Segmental; Breast Conserving Surgery; Cerenkov Luminescence Imaging; Beta particle detection
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Breast conserving surgery (Other): Females ≥ 30 years of age with a diagnosis of invasive breast cancer or ductal carcinoma in situ (DCIS), scheduled for BCS +/- SLNB or ALND
  Interventions: Device: EnLight; Device: LightPath

INTERVENTIONS:
Device: EnLight — The Lightpoint EnLight beta particle detector is an investigational non CE-marked medical device
Device: LightPath — The LightPath Imaging System is an investigational non CE-marked in vitro diagnostic device

SUMMARY:
This study will correlate the resection margin status of the breast cancer tumour (WLE specimen), cavity shavings (if any) and breast cavity, and the metastatic status of axillary lymph nodes as determined by EnLight, LightPath, and histopathology. This is a pilot study to assess feasibility before proceeding to a pivotal study to evaluate the use of these imaging systems in clinical practice.

DETAILED DESCRIPTION:
This is a prospective, single centre, pilot study to assess the feasibility of the EnLight and LightPath Imaging Systems for intra-operative analysis of tumour margins and axillary lymph nodes in breast conserving surgery (BCS) for breast cancer.

Female patients with a diagnosis of invasive breast cancer or DCIS scheduled to have BCS +/- sentinel lymph node biopsy (SLNB) or axillary lymph node dissection (ALND) will be screened, and enrolled in the study if eligible and willing to give written informed consent.

BCS only

Subjects scheduled to have BCS only will receive 5 MBq/kg of 18F-FDG, up to a maximum 300 MBq. 18F-FDG will be administered intravenously in the Nuclear Medicine Department, 60-180 minutes prior to EnLight and LightPath imaging.

After resection, the WLE specimen will be examined with the LightPath Imaging System. The WLE specimen will then be imaged with the EnLight Imaging System. The LightPath Imaging System will be located in a room next to the operating theatre, to allow "real-time" imaging to be performed. If a positive signal is detected with the EnLight Imaging System ("EnLight positive") or the LightPath Imaging System ("LightPath positive") the surgeon will perform cavity shavings of the positive area (up to a maximum thickness of 10mm). After resection, the shavings (if any) will be examined with the EnLight and LightPath Imaging Systems. A member of the research team who is not the operating surgeon will operate the LightPath Imaging System.

The EnLight will be used by the surgeon to image the surgical cavity post WLE. If the surgeon detects a positive signal with the EnLight, s/he will perform cavity shavings of the beta positive area (up to a maximum thickness of 10mm). All cavity shavings will be examined with the EnLight and LightPath Imaging Systems and then sent for histopathological analysis.

Sutures and/or surgical clips will be placed on the WLE specimen and cavity shavings (if performed) to record the anatomical orientation, as per standard practice. Positive signals on the resected WLE specimen and cavity shavings (if performed) will be marked by the surgeon with a prolene suture to facilitate accurate correlation with histopathology. If two or more positive signals are detected, multiple prolene sutures will be used.

BCS plus SLNB

Subjects scheduled to have BCS plus SLNB will receive 150 MBq 99mTc nanocolloid and 5 MBq/kg 18F-FDG, up to a maximum of 300 MBq. 99mTc nanocolloid will be injected periareolarly in the Nuclear Medicine Department prior to surgery. 18F-FDG will be administered intravenously in the Nuclear Medicine Department, 60-180 minutes prior to the estimated start of EnLight and LightPath imaging. The gamma probe will be used before and after the injection of 18F-FDG to identify and localise 99mTc SLN uptake transcutaneously. The findings before and after 18F-FDG injection will be compared to make sure 18F-FDG does not mask extraordinarily low active sentinel nodes. It is important to emphasize that we do not expect this to occur. Blue dye will be injected intra-operatively as per standard procedure.

BCS will be performed as described in section 'BCS only'.

As per standard practice the gamma probe and blue dye will be used to identify SLNs. Prior to dissection of the SLNs, the EnLight will be used by the surgeon to image the SLNs in vivo. All excised SLNs will be imaged with the EnLight and subsequently in the LightPath Imaging System at the time of the surgical procedure.

Following dissection of SLNs, the surgeon will scan the axilla with the EnLight to identify lymph nodes that are non-blue, non-palpable and gamma probe negative, but EnLight positive. EnLight positive lymph nodes will be excised and imaged with the EnLight and subsequently the LightPath Imaging System. As per SLNB standard of care the maximum number of lymph nodes that will be excised will be four in total.

The LightPath Imaging System will be located in a room next to the operating theatre, to allow "real-time" imaging to be performed. The EnLight positive and/or LightPath positive SLNs will be clearly labelled in order to facilitate correlation with histopathology.

BCS plus ALND

Subjects scheduled to have BCS plus ALND will receive 5 MBq/kg of 18F-FDG, up to a maximum 300 MBq. 18F-FDG will be administered intravenously in the Nuclear Medicine Department, 60-180 minutes prior to the estimated start of EnLight and LightPath imaging.

BCS will be performed as described in section 'BCS only'.

The surgeon will palpate the ALND specimen prior to complete resection to identify any palpable nodes. If present, palpable nodes will be imaged in vivo with the EnLight. The ALND specimen is then excised as per standard practice. The surgeon will examine the excised ALND tissue with the EnLight, and EnLight positive lymph nodes will be dissected from the ALND specimen. The maximum number of lymph nodes to be dissected from the ALND specimen will be four. All dissected lymph nodes will be imaged ex vivo with the EnLight and subsequently in the LightPath Imaging System at the time of the surgical procedure. The dissected lymph nodes will be sent separately for histopathological analysis to correlate the imaging findings with histopathology.

The LightPath Imaging Systems will be located in a room next to the operating theatre, to allow "real-time" imaging to be performed. The EnLight and/or LightPath positive SLNs will be clearly labeled in order to facilitate correlation with histopathology.

Histopathology of WLE specimen, shavings and lymph nodes

Following EnLight and LightPath imaging, the WLE specimen will be examined according to standard of care histopathology analysis. Details of tumour dimensions along with other histopathology minimum dataset items will be recorded. Additional sections of EnLight positive and/or LightPath positive areas that are marked with a prolene suture will be taken to facilitate accurate histopathology correlation. The additional sections will not affect standard of care histopathology analysis. The distance from the tumour to all six margins (medial, lateral, superior, inferior, anterior and posterior) will be recorded. A margin will be classified as positive if there is either invasive carcinoma within 1mm or DCIS within 2mm of the specimen surface as per current practice in the institution. Histopathology analysis will be performed on any tissue shavings obtained as a result of EnLight and/or LightPath imaging.

Lymph nodes will be examined according to standard of care histopathology analysis. The presence of any metastatic disease will be recorded and classified as macrometastasis (≥ 2 mm), micrometastasis (< 2 mm to > 0.2 mm) or isolated tumour cells (≤ 0.2 mm).

EnLight and LightPath imaging must be performed without unnecessary delay, and following the acquisition times set out in the IFU, in order to avoid any degradation in specimen quality prior to transfer to the tissue bank / pathology department for routine analyses.

Details of any adverse events will be recorded.

An ease of use questionnaire will be completed by the operators using the EnLight and LightPath, and by those interpreting recorded EnLight and LightPath images.

Radiation dosimetry

Staff in the Nuclear Medicine department will be monitored as per standard practice. Throughout the surgical procedure, all staff in the operating theatre will wear instant readout and monthly badge dosimeters. Staff handling the surgical specimens will also wear ring dosimeters. Staff caring for the subject in the recovery area will wear monthly badge dosimeters. Pathology staff processing the WLE and lymph node specimens will wear monthly badge and ring dosimeters.

Follow-up

Subject participation ends at the conclusion of the surgical procedure. Adverse events will be recorded until discharge, or for 24 hours after the first study procedure, whichever is sooner.

ELIGIBILITY:
Inclusion Criteria

Females ≥ 30 years of age with a diagnosis of invasive breast cancer or DCIS

Scheduled for BCS +/- SLNB or ALND

Females of childbearing age must have a negative pregnancy test (by Beta HCG qualitative analysis), must have a history of surgical sterilisation, or must give history of no menses in past twelve months

Exclusion Criteria

Surgery or radiotherapy in the operated breast in the past 2 years

Neoadjuvant systemic therapy

Patients not suitable for BCS

Blood glucose level ≥ 12 mmol/l on the day of surgery

Known hypersensitivity to 18F-FDG

Any patient who is pregnant or lactating

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-09; Primary Completion 2018-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility of intraoperative use of the EnLight and LightPath Imaging Systems. | Intra-operative
  The objective of this study is to assess the feasibility of the EnLight and LightPath Imaging Systems for intra-operative analysis of WLE specimens, the post-resection surgical cavity, shavings (if any) and axillary lymph nodes in vivo and ex vivo. This will be assessed by examining the following secondary outcome measures

SECONDARY OUTCOMES:
Tumour margin status of the WLE specimen (and shavings, if any) as determined by LightPath | Intra-operative

OTHER OUTCOMES:
Tumour margin status of the WLE specimen (and shavings, if any) as determined by EnLight | Intra-operatively
Tumour margin status of the post-resection breast surgical cavity as determined by EnLight | Intra-operatively
In vivo metastatic status of axillary lymph nodes as determined by EnLight | Intra-operatively
Ex vivo metastatic status of dissected lymph nodes as determined by EnLight | Intra-operatively
Ex vivo metastatic status of dissected lymph nodes as determined by the LightPath Imaging System | Intra-operatively
Radiation dosimetry to staff in the nuclear medicine department, operating theatre, recovery area and pathology lab | Peri-operatively
Ease of use | Peri-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Anand D Purushotham, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guy's Hospital, London, United Kingdom